CLINICAL TRIAL: NCT04942275
Title: Lung Perfusion PET / CT Using Gallium68-MMA for Preservation of Lung Function During Stereotactic Pulmonary Radiation Therapy
Brief Title: Lung Perfusion PET / CT Using Ga68-MAA for Preservation of Lung Function During Stereotactic Pulmonary Radiation Therapy
Acronym: PEGASUS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 29BRC21.0131
Record Dates: First submitted 2021-06-09; First posted 2021-06-28 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: SBRT; Non-small Cell Lung Cancer; Lung Metastasis
Keywords: Perfusion imaging; Positron EmissionTomography; Lung cancer; SBRT; Radiation induced lung injury
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention : Lung perfusion PET/CT using Ga68-MAA and SBRT planification (Experimental): All patients included for treatment with stereotactic radiotherapy for non-small cell lung cancer or lung metastasis will benefit from a pre-therapeutic functional assessment including:
  * The standard functional assessment recommended before performing an SBRT.
  * A perfusion PET/CT scan
  The treatment planning will be carried out in 2 stages:
  * First, an anatomical planning will be carried out, blinded to the PET results.
  * Then, a functional planning, respecting the standard constraints applied during anatomical planning, but also incorporating a new "functional lung volume" constraint defined by pulmonary PET, will then be carried out.
  A follow-up will be carried out for 12 months, including repeated perfusion PET/CT imaging at 3 and 12 months
  Interventions: Drug: Pre-therapeutic imaging test

INTERVENTIONS:
Drug: Pre-therapeutic imaging test — The radiopharmaceutical used for lung perfusion PET consists in human albumin macroaggregates labeled with Ga-68 (68Ga-MAA). 68Ga- MAA are administrated intravenously.

SUMMARY:
This is a prospective study evaluating the feasibility of treatment planning integrating lung perfusion PET/CT using Ga68-MAA to preserve functional lung areas during stereotactic body radiation therapy (SBRT).

DETAILED DESCRIPTION:
Lung perfusion PET / CT is a new imaging modality based on the use of the same cold molecules as those used for a conventional perfusion lung scan. Similartly, perfusion images are obtained after intravenous administration of human albumin macroaggregates, which are embolized in pulmonary capillaries according to pulmonary blood flow. However, these cold molecules are radiolabeled, not with Technetium99m, but with Gallium68, a ß + isotope, allowing image acquisition with PET technology. The same physiological processes are therefore observed with conventional scintigraphy PET imaging, but PET is an intrinsically superior technique for image acquisition, with greater sensitivity, better spatial and temporal resolutions and the possibility to perform respiratory-gated acquisition, allowing a better definition of the pulmonary functional volumes.

The aim is to evaluate the feasability of functional lung avoidance planification using lung perfusion PET/CT imaging during SBRT.

Patients will benefit from a pre-treatment functional assessment including PET/CT imaging.

The treatment planning will be carried out in 2 stages:

* First, an anatomical planning will be carried out, blinded to the PET results.
* Then, a functional planning, respecting the standard constraints applied during anatomical planning, but also incorporating a new "functional lung volume" constraint defined by PET/CT images, will be carried out.

A follow-up will be carried out for 12 months, including repeated perfusion PET/CT imaging at 3 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Insured patient
* Patient treated at the Brest CHRU for SBRT of a primary or secondary pulmonary lesion

Exclusion Criteria:

* Unable/unwilling to give informed consent
* Pregnancy / breast-feeding patient
* Patient under guardianship or curatorship
* Patient with contraindication to the administration of macroaggregates of human albumin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Patients with a dose reduction to the functional lung (estimated during functional planning). | Baseline, one week after lung perfusion PET / CT scan using Ga68-MAA
  Percentage of patients for whom it is possible to reduce the dose to the functional lung (estimated during the functional planning).
  A reduction in the dose to the functional lung will be defined by:
  * A decrease of at least 5% in functional lung volume included in V20Gy. or
  * A decrease of at least 5% in total relative lung function included in the V20G.

SECONDARY OUTCOMES:
Impact of lung perfusion PET / CT scan on lung activity during SBRT (stereotactic body radiation therapy) planning | Baseline, one week after lung perfusion PET / CT scan using Ga68-MAA
  Percentage of activity included in the V20Gy with the anatomical planning and the functional planning.
Impact of lung perfusion PET / CT scan on lung activity during SBRT (stereotactic body radiation therapy) planning | Baseline, one week after lung perfusion PET / CT scan using Ga68-MAA
  Percentage of functional lung volume included in the V20Gy with anatomical planning and during functional planning
Pulmonary toxicity at 3 months | At 3 months after SBRT (stereotactic body radiation therapy)
  Pulmonary toxicity defined according to EORTC (European Organisation for Research and Treatment of Cancer) criteria (Common Terminology Criteria for Adverse Events 5.0, EORTC QLQ-C30 : European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire - Cancer module 30) at 3 months
Pulmonary toxicity at 3 months | At 3 months after SBRT( stereotactic body radiation therapy)
  Pulmonary toxicity defined according to EORTC (European Organisation for Research and Treatment of Cancer) criteria (Common Terminology Criteria for Adverse Events 5.0, EORTC QLQ-LC13 :European Organisation for Research and Treatment of Cancer- Quality of Life Questionnaire - Lung Cancer module 13) at 3 months
Pulmonary toxicity at 6 months | At 6 months after SBRT (stereotactic body radiation therapy)
  Pulmonary toxicity defined according to EORTC (European Organisation for Research and Treatment of Cancer) criteria (Common Terminology Criteria for Adverse Events 5.0, EORTC QLQ-C30 : European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire -Cancer module 30) at 6 months
Pulmonary toxicity at 6 months | At 6 months after SBRT (stereotactic body radiation therapy)
  Pulmonary toxicity defined according to EORTC (European Organisation for Research and Treatment of Cancer) criteria (Common Terminology Criteria for Adverse Events 5.0, EORTC QLQ-LC13 : European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire - Lung Cancer module 13) at 6 months
Pulmonary toxicity at 9 months | At 9 months after SBRT (stereotactic body radiation therapy)
  Pulmonary toxicity defined according to EORTC (European Organisation for Research and Treatment of Cancer) criteria (Common Terminology Criteria for Adverse Events 5.0, EORTC QLQ-C30 : European Organisation for Research and Treatment of Cancer -Quality of Life Questionnaire - Cancer module 30) at 9 months
Pulmonary toxicity at 9 months | At 9 months after SBRT (stereotactic body radiation therapy)
  Pulmonary toxicity defined according to EORTC (European Organisation for Research and Treatment of Cancer) criteria (Common Terminology Criteria for Adverse Events 5.0, EORTC QLQ-LC13 : European Organisation for Research and Treatment of Cancer -Quality of Life Questionnaire - Lung Cancer module 13) at 9 months
Pulmonary toxicity at 12 months | At 12 months after SBRT (stereotactic body radiation therapy)
  Pulmonary toxicity defined according to EORTC (European Organisation for Research and Treatment of Cancer) criteria (Common Terminology Criteria for Adverse Events 5.0, EORTC QLQ-C30 : European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire - Cancer module 30) at 12 months
Pulmonary toxicity at 12 months | At 12 months after SBRT (stereotactic body radiation therapy)
  Pulmonary toxicity defined according to EORTC (European Organisation for Research and Treatment of Cancer) criteria (Common Terminology Criteria for Adverse Events 5.0, EORTC QLQ-LC13 : European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire - Lung Cancer module 13) at 12 months
Dyspnea at Day 0 (inclusion) | Baseline, Day 0
  Results of EuroQol (EQ-5D-5L) questionnaire
Dyspnea at Day 0 (inclusion) | Baseline, Day 0
  Results of Pulmonary Function testing (PFT) : FEV1
Dyspnea at Day 0 (inclusion) | Baseline, Day 0
  Results of Pulmonary Function testing (PFT) : FEV1/FVC
Dyspnea at Day 0 (inclusion) | Baseline, Day 0
  Results of 6 minutes Walk Test (6MWT)
Dyspnea at 3 months | At 3 months after SBRT (stereotactic body radiation therapy)
  Results of EuroQol (EQ-5D-5L) questionnaire
Dyspnea at 3 months | At 3 months after SBRT (stereotactic body radiation therapy)
  Results of Pulmonary Function testing (PFT) : FEV1
Dyspnea at 3 months | At 3 months after SBRT (stereotactic body radiation therapy)
  Results of Pulmonary Function testing (PFT) : FEV1/FVC
Dyspnea at 3 months | At 3 months after SBRT (stereotactic body radiation therapy)
  Results of 6 minutes Walk Test (6MWT)
Dyspnea at 6 months | At 6 months after SBRT (stereotactic body radiation therapy)
  Results of EuroQol (EQ-5D-5L) questionnaire
Dyspnea at 6 months | At 6 months after SBRT (stereotactic body radiation therapy)
  Results of Pulmonary Function testing (PFT) : FEV1
Dyspnea at 6 months | At 6 months after SBRT (stereotactic body radiation therapy)
  Results of Pulmonary Function testing (PFT) : FEV1/FVC
Dyspnea at 6 months | At 6 months after SBRT (stereotactic body radiation therapy)
  Results of 6 minutes Walk Test (6MWT)
Dyspnea at 9 months | At 9 months after SBRT (stereotactic body radiation therapy)
  Results of EuroQol (EQ-5D-5L) questionnaire
Dyspnea at 9 months | At 9 months after SBRT (stereotactic body radiation therapy)
  Results of Pulmonary Function testing (PFT) : FEV1
Dyspnea at 9 months | At 9 months after SBRT (stereotactic body radiation therapy)
  Results of Pulmonary Function testing (PFT) : FEV1/FVC
Dyspnea at 9 months | At 9 months after SBRT (stereotactic body radiation therapy)
  Results of 6 minutes Walk Test (6MWT)
Dyspnea at 12 months | At 12 months after SBRT (stereotactic body radiation therapy)
  Results of EuroQol (EQ-5D-5L) questionnaire
Dyspnea at 12 months | At 12 months after SBRT (stereotactic body radiation therapy)
  Results of Pulmonary Function testing (PFT) : FEV1
Dyspnea at 12 months | At 12 months after SBRT (stereotactic body radiation therapy)
  Results of Pulmonary Function testing (PFT) : FEV1/FVC
Dyspnea at 12 months | At 12 months after SBRT (stereotactic body radiation therapy)
  Results of 6 minutes Walk Test (6MWT)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, Brest Cedex, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Le Roux PY, Le Pennec R, Bourbonne V, Blanc-Beguin F, Pavoine M, Kerleguer K, Mauguen M, Pradier O, Salaun PY, Lucia F, Bourhis D. Pulmonary uptake value (PUV): a new quantification method for lung PET/CT imaging. EJNMMI Res. 2025 Jul 1;15(1):79. doi: 10.1186/s13550-025-01274-y. PMID 40591115